CLINICAL TRIAL: NCT01796015
Title: Intracranial Hypertension Detection Using Optic Nerve Sheath Diameter Measurement in Children
Brief Title: Intracranial Hypertension and Optic Nerve Sheath Diameter
Acronym: DENO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010.598; 2010-A00890-39 (Other: ID-RCB)
Record Dates: First submitted 2012-10-25; First posted 2013-02-21 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Cerebral Stroke; Cerebral Venous Thrombosis
Keywords: paediatrics; optic nerve sheath diameter; ultrasound
MeSH Terms: conditions — Stroke; Intracranial Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- For the 97 patients (Other): * day 0: ultrasound of ONSD (= 4 measurements: 1 transverse and 1 sagittal for each eye) + transcranial Doppler at T-15 (15 minutes before ICP measurement), within 1h following ICP measurement, and one more measurement is to be done if significant ICP variations are noticed (variation over 15 mmHg during at least 5 minutes)
  * day 1: ONSD ultrasound + transcranial Doppler in the morning and one more measurement is to be done if significant ICP variations are noticed (variation over 15 mmHg during at least 5 minutes)
  * days 2 and 3 : same as day 1
  * when leaving the intensive care unit: Pediatric Overall Performance Category (POPC) scale
  Interventions: Other: ONSD ultrasound
- For the control group (Other): one single ONSD in addition to their usual care (4 measurements: 1 transverse and 1 sagittal for each eye) in the morning in absence of painful sensation
  Interventions: Other: ONSD ultrasound
- For the learning curve (Other): minimum 15 ONSD ultrasounds will be performed by each of the 15 intensive care doctor or interns expected. One ONSD ultrasound corresponds to 2 measurements: 1 transverse and 1 sagittal. Each volunteer will have maximum 30 ONSD ultrasound measures over a 1 month period.
  Interventions: Other: ONSD ultrasound

INTERVENTIONS:
Other: ONSD ultrasound — Description of the ONSD ultrasound: ONSD is measured 3 mm behind the globe and perpendicularly to the optic nerve axis (2 dimensions mode).
  For each optic nerve, 2 measures are performed: 1 sagittal and 1 transverse. The patient is positioned in 30° dorsal elevation. Gel is applied on the eyelid and a 7,5 MHz probe is used.
  At the same time and on the same side, a transcranial Doppler is performed using a 2 MHz probe placed on the temple. Are measured: systolic velocity, mean velocity, diastolic velocity, resistance index and pulsatility index.
  As ONSD measures cannot be done blinded (regarding ICP monitoring), a centralised evaluation (by 2 experts) of the recorded sonograms is planned.

SUMMARY:
Intracranial hypertension (ICH) is a mortality risk factor in severe traumatic brain injury (TBI), in purulent meningitis, in hepatic encephalopathy and in Reye's syndrome. It is also a risk factor for severe neurologic sequelae in survivors. Intracranial pressure (ICP) monitoring is likely to guide therapeutics, and certain research on adults or on children, suggest that IH therapeutic approach, for instance for bacterial meningitis, would improve the prognosis. Two monitoring techniques are currently recommended. They are reference methods for ICP measure :

* monitoring with intraventricular catheter,
* intra-parenchymal monitoring using optical fiber catheter. Non invasive methods have been suggested, including ultrasound measurement of optic nerve sheath diameter (ONSD) which is the most interesting one. The ONSD measured ultrasonically is correlated with ICP level in adults with severe TBI. A diameter over 5,9 mm predicts ICH within the first 24 hours. In children, ONSD average values have been worked out, and an ONSD increase is found in children suffering from hydrocephalus with IH and in children with TBI. ICH precocious detection is fundamental in children sensitive to ICH because their cerebral development is not finished yet. Difficulties met for ICP monitoring implementation in infants and its invasive nature are often disliked by clinicians. A non-invasive exam is then essential to allow a better care of children with ICH in intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

For the 97 patients:

* children from 2 months to 16 years
* in the intensive care unit
* TBI : moderate (GCS between 9 and 12) to severe (GCS <9), whatever the mechanism involved
* informed consent form signed by parents

Non inclusion Criteria:

* obesity (BMI > 97th percentile for the age)
* patient already under replacement therapy.
* patient taking AEDs
* patient with long-term systemic corticosteroid therapy
* history of neurological disease or learning difficulties
* no covered by a national health insurance

Ages: 2 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2011-04; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Primary (sensitivity and specificity of echographic measurement of ONSD) | To determine diagnostic performance (sensitivity and specificity) of ICH thanks to ultrasound measurement of ONSD, (15 minutes ,before invasive ICP monitoring)
  Sensitivity and specificity of echographic measurement of the ONSD (mean value of both eyes), taken 15 minutes ,before invasive ICP monitoring, regarding detection of ICH in children with neurological injury, as compared to reference method for ICH detection (ICP monitoring with intraventricular catheter).

SECONDARY OUTCOMES:
Secondary outcome (1. To draw learning curves before the study begins to find out the number of ultrasound measurement needed) | 1. To draw learning curves before the study begins to find out the number of ultrasound measurement needed (day 0)
  * value (mm) of the echographic ONSD measurement performed by the clinicians/interns (learning curve) compared to the value found by the trainer
  * mean value, standard deviation and quartiles of ONSD measures performed in a population of patients intubated, ventilated, sedated and without cerebral lesion (control group)
  * Correlation between echographic ONSD values (mean of the values) and invasive ICP monitoring values (taken same day)
  * Correlation between variations of ONSD measures and treatment effet on ICH
  * Comparison of diagnostic capacity of ONSD measurements depending on age, ICH etiology (bacterial meningitis, encephalitis meningitis, stroke, cerebral cerebral thrombophlebitis, TBI and patients from neurosurgery)
  * determine diagnostic capacity of the measures performed with transcranial Doppler (resistance index, pulsatility index, systolic, mean and diastolic velocities) in the different pathologies and compare them to ONSD values

CONTACTS AND LOCATIONS:
Overall Officials: Etienne JAVOUHEY, MD, Principal Investigator — HOPITAL FEMME MERE ENFANT HOSPICES CIVILS DE LYON
Locations (2):
- France (2):
  - Pediatric Critical Care Unit, Hôpital Femme Mère Enfant ,Hospices Civils de Lyon, Bron, Auvergne-Rhône-Alpes
  - Pediatric Critical Care Unit, CHU La Tronche, Grenoble

REFERENCES:
- [Result] Cour-Andlauer F, Portefaix A, Wroblewski I, Rabilloud M, Bordet F, Cogniat B, Didier C, Pouyau R, Valla FV, Kassai-Koupai B, Simeon G, Ginhoux T, Courtil-Teyssedre S, Javouhey E. Predictive Value of Optic Nerve Sheath Diameter for Diagnosis of Intracranial Hypertension in Children With Severe Brain Injury. Front Pediatr. 2022 Jun 6;10:894449. doi: 10.3389/fped.2022.894449. eCollection 2022. PMID 35733810